CLINICAL TRIAL: NCT01106989
Title: An Open-label Pilot Study Evaluating Synera® in the Treatment of Patients With Pain Associated With Myofascial Trigger Points
Brief Title: Study Evaluating Heated Lidocaine/Tetracaine Patch in Patients With Pain Associated With Myofascial Trigger Points
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ZARS Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SC-203
Record Dates: First submitted 2010-04-16; First posted 2010-04-20 (Estimated); Last update posted 2012-03-16 (Estimated); Status verified 2012-03

CONDITIONS: Myofascial Pain Syndromes
MeSH Terms: conditions — Myofascial Pain Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Heated lidocaine/tetracaine patch (Experimental): Active
  Interventions: Drug: Heated lidocaine/tetracaine patch

INTERVENTIONS:
Drug: Heated lidocaine/tetracaine patch — Patients will be instructed to apply one heated lidocaine 70 mg and tetracaine 70 mg topical patch directly to each trigger point identified at the Screening/Baseline Visit (up to 3 trigger points). Patches will be administered for 4 hours, 2 times per day (total of 8 hours for each trigger point per day).
  Other Names: Synera

SUMMARY:
The purpose of this pilot study is to explore the potential usefulness of a heated lidocaine 70 mg and tetracaine 70 mg topical patch for the treatment of pain associated with myofascial trigger points.

DETAILED DESCRIPTION:
The purpose of this pilot study is to explore the usefulness of a heated lidocaine 70 mg and tetracaine 70 mg topical patch for the treatment of pain associated with myofascial trigger points. The study will consist of a 2-week, open-label treatment period followed by a 2 week follow-up period conducted at a single study site. Eligible patients must have a clinical diagnosis of pain (minimum 1-month duration) associated with up to 3 identifiable myofascial trigger points. A number of efficacy variables will be employed to evaluate their utility for assessing painful responses in this population.

ELIGIBILITY:
Inclusion Criteria:

* be at least 18 years of age
* have a clinical diagnosis of pain (minimum 1-month duration) associated with up to 3 myofascial trigger points
* have trigger points confined to the upper back, shoulder, and neck

Exclusion Criteria:

* have used any topically applied pain medication on the target treatment area within 3 days preceding the Screening/Baseline Visit
* have used any topically applied pain medication on the target treatment area within 3 days preceding the Screening/Baseline Visit
* have used any injected pain medication with 28 days preceding the Screening/Baseline Visit
* are receiving class 1 antiarrhythmic drugs (ie, tocainide, mexiletine, etc.)

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-06; Primary Completion 2010-12 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Pain intensity | Two weeks

SECONDARY OUTCOMES:
Pain interference with activities (eg, general, normal work, sleep) | Two weeks

CONTACTS AND LOCATIONS:
Overall Officials: Richard L Rauck, MD, Principal Investigator — The Center for Clinical Research
Locations (1):
- The Center for Clinical Research, Winston-Salem, North Carolina, United States